CLINICAL TRIAL: NCT00326664
Title: A Phase I Clinical Trial of AZD2171 in Children With Recurrent or Progressive Central Nervous System (CNS) Tumors
Brief Title: AZD2171 in Treating Young Patients With Recurrent, Progressive, or Refractory Primary CNS Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00709; NCI-2009-00709 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000476579; PBTC-020; PBTC-020 (Other: Pediatric Brain Tumor Consortium); PBTC-020 (Other: CTEP); U01CA081457 (NIH)
Record Dates: First submitted 2006-05-16; First posted 2006-05-17 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-03

CONDITIONS: Childhood Atypical Teratoid/Rhabdoid Tumor; Childhood Central Nervous System Germ Cell Tumor; Childhood Cerebral Anaplastic Astrocytoma; Childhood Cerebral Astrocytoma; Childhood Grade I Meningioma; Childhood Grade II Meningioma; Childhood Grade III Meningioma; Childhood Infratentorial Ependymoma; Childhood Oligodendroglioma; Childhood Spinal Cord Neoplasm; Childhood Supratentorial Ependymoma; Recurrent Childhood Brain Neoplasm; Recurrent Childhood Brain Stem Glioma; Recurrent Childhood Cerebellar Astrocytoma; Recurrent Childhood Cerebral Astrocytoma; Recurrent Childhood Ependymoma; Recurrent Childhood Medulloblastoma; Recurrent Childhood Pineoblastoma; Recurrent Childhood Subependymal Giant Cell Astrocytoma; Recurrent Childhood Supratentorial Primitive Neuroectodermal Tumor; Recurrent Childhood Visual Pathway Glioma
MeSH Terms: conditions — Rhabdoid Tumor; Astrocytoma; Oligodendroglioma; Spinal Cord Neoplasms; Familial ependymoma; Medulloblastoma; Optic Nerve Glioma | interventions — cediranib

ARMS (1):
- Treatment (cediranib maleate) (Experimental): Patients receive oral AZD2171 once daily on days 1-28. Treatment repeats every 28 days for up to 13 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cediranib Maleate

INTERVENTIONS:
Drug: Cediranib Maleate — Given orally
  Other Names: AZD2171; AZD2171 Maleate; Recentin

SUMMARY:
This phase I trial is studying the side effects and best dose of AZD2171 in treating young patients with recurrent, progressive, or refractory primary CNS tumors. AZD2171 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose of AZD2171 in pediatric patients with recurrent, progressive, or refractory primary CNS tumors.

II. Describe the toxicity profile and dose-limiting toxicities of AZD2171 in these patients.

SECONDARY OBJECTIVES:

I. Characterize inter-patient variability in the pharmacokinetics of AZD2171 in these patients.

II. Describe changes in circulating endothelial cells (CECs) and circulating endothelial cell precursors (CEPs) in patients treated with AZD2171 at different dose levels.

III. Correlate changes in CECs, CEPs, plasma, serum, and urine levels of proteins with angiogenesis, including vascular endothelial growth factor (VEGF) and VEGF receptor, in patients treated with AZD2171 at different dose levels.

IV. Correlate changes in CECs, CEPs, and angiogenic modulators with changes in magnetic resonance (MR) perfusion.

V. Obtain preliminary evidence of biologic activity of AZD2171 by evaluating alterations in tissue perfusion, tumor blood flow, and metabolic activity using MR perfusion and diffusion imaging, and positron-emission tomography, and correlating these findings with changes in tumor size by standard MRI.

OUTLINE: This is a dose-escalation, multicenter study. Patients are stratified according to concurrent enzyme-inducing anticonvulsant drugs (yes vs no).

Patients receive oral AZD2171 once daily on days 1-28. Treatment repeats every 28 days for up to 13 courses in the absence of disease progression or unacceptable toxicity.

For each stratum, cohorts of 2-6 patients receive escalating doses of AZD2171 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 25% of patients experience dose-limiting toxicity. Once the MTD is determined, an additional 6 patients per stratum are enrolled and treated at the MTD.

After completion of study, patients are followed at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary CNS tumor

  * Histologically benign brain tumors (e.g., low-grade glioma) allowed
  * Histological requirement waived for intrinsic brain stem or diffuse optic pathway tumors, but must have clinical and/or radiographic evidence of progression
* Recurrent, progressive, or refractory disease
* Absolute neutrophil count >= 1,000/mm^3 (unsupported)
* Platelet count >= 75,000/mm^3 (unsupported)
* Creatinine =< 1.5 times upper limit of normal (ULN) OR glomerular filtration rate >= 70 mL/min
* Bilirubin =< 1.5 times ULN
* ALT =< 2.5 times ULN
* Urine dipstick or urinalysis < 1+ protein
* Albumin >= 3 g/dL
* Karnofsky performance status (PS) 60-100% (> 16 years of age) OR Lansky PS 60-100% (=< 16 years of age)
* Karnofsky/Lansky PS 70-100% for patients at increased risk for compromised LVEF
* Hemoglobin >= 8 g/dL (transfusion support allowed)
* No overt renal, hepatic, cardiac, or pulmonary disease
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* QTc prolongation =< 500 msec
* No other significant ECG abnormality within the past 14 days
* No clinically significant, unrelated, systemic illness, including serious infections or significant cardiac, pulmonary, hepatic, or other organ dysfunction, that would preclude study participation
* No uncontrolled hypertension

  * Defined as systolic and diastolic BP > 95th percentile for age (ages 1-17)
  * Defined as BP > 140/90 (ages 18 and older)
* No New York Heart Association class III or IV disease and Karnofsky/Lansky PS < 70

  * Class II disease controlled with treatment and increased monitoring is allowed
* Recovered from all prior therapy
* No prior AZD2171
* At least 3 weeks since prior myelosuppressive anticancer chemotherapy (6 weeks for nitrosoureas)
* More than 1 weeks since prior investigational or biologic agents

  * If the investigational or biologic agent has a prolonged half-life (> 48 hours), then these patients must be discussed with the study chair prior to registration
* No concurrent drugs or biologics with proarrhythmic potential
* More than 3 months since last fraction of craniospinal radiotherapy or total-body irradiation
* More than 4 weeks since last fraction of focal irradiation to symptomatic metastatic sites
* At least 6 months since prior allogeneic bone marrow transplantation
* At least 3 months since prior autologous bone marrow or stem cell transplantation
* At least 1 week since prior filgrastim (G-CSF), sargramostim (GM-CSF), or epoetin alfa (2 weeks for pegfilgrastim)
* No other concurrent investigational agents
* Concurrent dexamethasone allowed provided patient is on a stable or decreasing dose for ≥ 1 week before study entry
* No concurrent chemotherapy
* No concurrent routine use of G-CSF, GM-CSF, or epoetin alfa
* Able to swallow tablets
* Any neurologic deficits must be stable for >= 1 week
* If the investigational or biologic agent has a prolonged half-life (> 48 hours), then these patients must be discussed with the study chair prior to registration

Exclusion Criteria:

* No known curative therapy available

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 55 (Actual)
Dates: Start 2006-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose, defined as the dose at which the model estimates that 25% of patients will experience dose-limiting toxicity as measured by NCI CTCAE v4.0 | 42 days
  Estimated using the modified Continual Reassessment Method (CRM).

CONTACTS AND LOCATIONS:
Overall Officials: Mark Kieran, Principal Investigator — Pediatric Brain Tumor Consortium
Locations (11):
- United States (11):
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Dana-Farber/Harvard Cancer Center, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Pediatric Brain Tumor Consortium, Memphis, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington